CLINICAL TRIAL: NCT06732245
Title: A Randomized, Double-Blind, Placebo-Controlled Multi-Center Study of Oral NA-931, Alone or in Addition to Open Label Subcutaneous Tirzepatide , to Investigate the Efficacy and Safety in Overweight or Obese Men and Women
Brief Title: Safety and Efficacy of NA-931 and Tirzepatide in Adults Who Are Overweight or Obese
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biomed Industries, Inc. (Industry)
Collaborators: Bioneurals Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NA-931-200
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: NA-931; Obesity; Biomed Industries, Inc; overweight; Tirzepatide; Zepbound
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: The study is designed to have three periods. The 48-week core treatment period has 9 treatment arms, with combinations of 3 Tirzepatide doses (none, 2.5 mg and 5 mg and 10 mg injectable) and 3 NA-931 doses (0, 60 mg and 150 mg oral). The core treatment period is then followed by an open-label 12-week treatment extension period during which participants originally assigned to either placebo or NA-931 60 mg will switch to NA-931 150 mg. All other treatment assignments will remain the same. The extension period is then followed by a 12-week post-treatment period, during which all study treatments will be withdrawn from all arms.
Who Masked: Participant, Investigator
Masking Description: With regards to NA-931 and placebo-NA-931, the participants, Investigator and Sponsor will be blinded.
  Due to Tirzepatide being pre-filled, packaged and labeled by manufacturer, it is not possible to blind Tirzepatide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Placebo Comparator: Placebo (Placebo Comparator): Placebo Comparator: Placebo to oral NA-931 120 mg daily + no Tirzepatide Participants will receive oral placebo at baseline and at Weeks 4, 12, and 24, 36, and 48 during the core treatment period and will switch during the extension period to receive NA-931 60 mg daily at Weeks 60 and 72.
  Interventions: Drug: NA-931
- Placebo + Tirzepatide 5 mg (Placebo Comparator): Other: Placebo + Tirzepatide 5 mg Participants will receive oral placebo at baseline and at Weeks 4, 12, and 24, 36, and 48, and s.c. Tirzepatide 5 mg weekly per the dose escalation schedule.
  Interventions: Drug: NA-931
- Placebo + Tirzepatide 10 mg (Placebo Comparator): Placebo + Tirzepatide 10 mg Participants will receive oral placebo at baseline and at Weeks 4, 12, and 24, 36, and 48 and s.c. Tirzepatide 10 mg weekly per the dose escalation schedule.
  Interventions: Drug: NA-931 150 mg + no Tirzepatide
- NA-931 60mg to NA-931 150 mg + no Tirzepatide (Experimental): Experimental: NA-931 60mg to NA-931 150 mg + no Tirzepatide Participants will receive oral NA-931 60 mg at baseline and at Weeks 4, 12, and 24, 36, and 48 during the core treatment period and will switch during the extension period to receive NA-931 60 mg at Weeks 60 and 72.
  Interventions: Drug: NA-931
- NA-931 60 mg + Tirzepatide 5 mg (Active Comparator): NA-931 60 mg + Tirzepatide 5 mg Participants will receive oral NA-931 60 mg at baseline and at Weeks 4, 12, and 24, 36, and 48 and s.c. Tirzepatide 5 mg weekly per the dose escalation schedule.
  Interventions: Drug: NA-931
- NA-931 120 mg + Tirzepatide 5 mg (Active Comparator): NA-931 120 mg + Tirzepatide 5 mg Participants will receive oral NA-931 60 mg at baseline and at Weeks 4, 12, and 24, 36, and 48 and s.c. Tirzepatide 5 mg weekly per the dose escalation schedule.
  Interventions: Drug: NA-931
- NA-931 150 mg + no Tirzepatide (Experimental): Experimental: NA-931 150 mg + no Tirzepatide Participants will receive oral NA-931 150 mg at baseline and at Weeks 4, 12, 24, 36 and 48
  Interventions: Drug: Tirzepatide
- NA-931 150 mg + Tirzepatide 2.5 mg (Active Comparator): NA-931 150 mg + Tirzepatide 2.5 mg Participants will receive oral NA-931 150 mg at baseline, and at Weeks 4, 12, and 24, 36, and 48 and s.c. Tirzepatide 2.5 mg weekly per the dose escalation schedule.
  Interventions: Drug: Tirzepatide
- NA-931 150 mg + Tirzepatide 5 mg (Active Comparator): NA-931 150 mg + Tirzepatide 5 mg Participants will receive oral NA-931 150mg at baseline and at Weeks 4, 12, and 24, 36, and 48 and s.c. Tirzepatide 5 mg per the dose escalation schedule.
  Interventions: Drug: NA-931

INTERVENTIONS:
Drug: NA-931 — NA-931 (oral, daily), a quadruple receptor agonist
  Tirzepatide (Zepbound) placebo
  Other Names: Tirzepatide placebo
  Arms: NA-931 120 mg + Tirzepatide 5 mg
Drug: Tirzepatide — Tirzepatide (s.c. weekly)
  * Glucagon-like peptide-1 (GLP-1) receptor agonist
  * Other Names:
    * Mounjaro
    * Zepbound NA-931 Placebo (oral, daily)
  Other Names: NA-931 Placebo
  Arms: NA-931 150 mg + no Tirzepatide
Drug: Tirzepatide — Tirzepatide (s.c. weekly), a Glucagon-like peptide-1 (GLP-1) receptor agonist
  • Other Names:
  * Mounjaro
  * Zepbound
  NA-931 Placebo (oral, daily)
  Other Names: NA-931 Placebo
  Arms: NA-931 150 mg + Tirzepatide 2.5 mg
Drug: NA-931 — NA-931, an oral, daily
  • A quadruple receptor agonist
  Arms: NA-931 150 mg + Tirzepatide 5 mg
Drug: NA-931 — NA-931 (oral, daily), a quadruple receptor agonist
  Tirzepatide (s.c. weekly)
  * Glucagon-like peptide-1 (GLP-1) receptor agonist
  * Other Names:
    * Mounjaro
    * Zepbound
  Other Names: Tirzepatide
  Arms: NA-931 60 mg + Tirzepatide 5 mg
Drug: NA-931 — NA-931 (oral daily), a quadruple receptor agonist
  Tirzepatide (s.c. weekly)
  * Glucagon-like peptide-1 (GLP-1) receptor agonist
  * Other Names:
    * Mounjaro
    * Zepbound
  Other Names: Tirzepatide
  Arms: NA-931 60mg to NA-931 150 mg + no Tirzepatide
Drug: NA-931 150 mg + no Tirzepatide — NA-931 150 mg + no Tirzepatide
  Arms: Placebo + Tirzepatide 10 mg
Drug: NA-931 — NA-931 (oral, daily), a quadruple receptor agonist
  Tirzepatide (s.c. weekly)
  * Glucagon-like peptide-1 (GLP-1) receptor agonist
  * Other Names:
    * Mounjaro
    * Zepbound
  Other Names: Tirzepatide
  Arms: Placebo + Tirzepatide 5 mg
Drug: NA-931 — NA-931 (oral, daily), a quadruple receptor agonist
  Tirzepatide (s.c. weekly)
  * Glucagon-like peptide-1 (GLP-1) receptor agonist
  * Other Names:
    * Mounjaro
    * Zepbound
  Other Names: Tirzepatide
  Arms: Placebo Comparator: Placebo

SUMMARY:
A phase 2 study to assess the efficacy of NA-931 alone or in addition to Tirzepatide to assess efficacy and safety in overweight or obese men and women

DETAILED DESCRIPTION:
This Phase 2 study investigates if NA-931 in addition to Tirzepatide can demonstrate synergic effects by enhancing efficacy and reducing adverse events including preserve/increase muscle mass in the presence of weight and/or fat mass loss.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent must be obtained before any study-related assessments are performed.
* Men and women between 18 and 80 years, inclusive; women of child-bearing potential (defined as those who are not post-menopausal or post-surgical sterilization) must meet both of the following criteria:

  * Two negative pregnancy tests (at screening and at randomization, prior to dosing)
  * Use of intrauterine device, from at least 3 months before the baseline visit through at least 4 months after the last dose of NA-931/placebo oral, and an additional contraceptive (barrier) method from screening through at least 4 months after the last dose of NA-931/placebo oral.
* Body mass index (BMI) ≥ 30 or BMI ≥ 27 with one or more obesity-associated comorbidities (e.g., hypertension, insulin resistance, sleep apnea, or dyslipidemia)
* Stable body weight (± 5 kg) within 90 days of screening, and body weight <150 kg
* Have a history of at least one self-reported unsuccessful behavioral effort to lose body weight
* Able to communicate well with the Investigator, comply with the study requirements and adhere to the diet and activity programs for the study duration

Exclusion Criteria:

* • History of, or known hypersensitivity to, monoclonal antibody drugs or a contraindication to Tirzepatide (Zepbound® or Mounjaro®)

  * Use of other investigational drugs at the time of enrollment or within 30 days or 5 half-lives of enrollment, whichever is longer, or longer if required by local regulations
  * Treatment with any medication for the indication of obesity within the past 30 days before screening
  * Diagnosis of diabetes requiring current use of any antidiabetic drug or HbA1c ≥ 6.5% Note: Metabolic syndrome is not an exclusion, even if managed with an anti-diabetic drug such as metformin or an SGLT2 inhibitor. A diagnosis of prediabetes or impaired glucose tolerance managed exclusively with non-pharmacologic approaches (e.g., diet and exercise) is not an exclusion.
  * Any chronic infections likely to interfere with study conduct or interpretation such as hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV). History of hepatitis A or hepatitis C successfully treated is not exclusionary. Active COVID-19 infection.
  * Donation or loss of 400 mL or more of blood within 8 weeks prior to initial dosing, or longer if required by local regulation, or plasma donation (> 250 mL) within 14 days prior to the first dose
  * Any disorder, unwillingness, or inability not covered by any of the other exclusion criteria, which in the Investigator's opinion, might jeopardize the participant's safety or compliance with the protocol

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight at 48 weeks | 48 weeks
  Change in total body weight will be measured from baseline to 48 weeks

SECONDARY OUTCOMES:
Change from baseline in waist circumference (cm) at 48 weeks | 48 weeks
  Waist circumference will be measured in standing position with a non-stretchable measuring tape and to the nearest 0.1 centimeter (cm).
Change from baseline at 48 weeks in total body fat mass in kilograms (kg) | 48 weeks
  Fat mass will be obtained by dual-energy x-ray absorptiometry (DXA) Dual energy X-ray absorptiometry (DXA) will be used to assess changes in body composition.
Change from baseline at 48 weeks in percent body fat | 48 weeks
  Percent body fat will be obtained by dual-energy x-ray absorptiometry (DXA) Dual energy X-ray absorptiometry (DXA) will be used to assess changes in body composition.
Change from baseline at 48 weeks in visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and trunk fat mass by dual-energy x-ray absorptiometry (DXA) | 48 weeks
  Dual energy X-ray absorptiometry (DXA) will be used to assess changes in body composition.
Proportion of participants at 48 weeks with change in waist circumference ≥ 5 cm | 48 weeks
  Waist circumference will be measured in standing position with a non-stretchable measuring tape and to the nearest 0.1 centimeter (cm).
Proportion of participants at 48 weeks with change in Body weight ≥ 5%, ≥ 10% and ≥15% | 48 weeks
  Body weight will be measured in kilograms (kg) to the nearest 0.1 kg.
Proportion of participants at 48 weeks with change in Fat mass ≥ 5% ≥ 10% ≥ 15% by Dual energy X-ray absorptiometry (DXA) | 48 weeks
  Dual energy X-ray absorptiometry (DXA) will be used to assess the changes in body composition.
Proportion of participants at 48 weeks with change in Fat mass ≥ 10% with <5% decrease (or and increase) in lean mass by Dual energy X-ray absorptiometry (DXA) | 48 weeks
  Dual energy X-ray absorptiometry (DXA) will be used to assess changes in body composition.
Percentage of weight loss due to fat mass or lean mass at 48 weeks by dual-energy x-ray absorptiometry (DXA) | 48 weeks
  Dual energy X-ray absorptiometry (DXA) will be used to assess changes in body composition
Change from baseline at 48 weeks in fat mass (kg and %) by bioelectrical impedance analysis (BIA) | 48 weeks
  Bioelectrical impedance analysis (BIA) is a widely used method for estimating body composition.
Change from baseline at 48 weeks in lean mass (kg and %) and appendicular lean mass by dual-energy x-ray absorptiometry (DXA) | 48 weeks
  Dual-energy x-ray absorptiometry (DXA) will be used to assess changes in body composition.
Change from baseline at 48 weeks in lean mass (kg) by bioelectrical impedance analysis (BIA) | 48 weeks
  Bioelectrical impedance analysis (BIA) is a widely used method for estimating body composition.
Safety and tolerability measurements throughout 48 weeks by TEAEs [safety labs, vital signs] | 48 weeks
  Incidence and severity of treatment emergent adverse events (TEAEs)
Proportion of Participants with change from baseline in Body Mass Index (BMI) categories at 48 weeks | 48 weeks
  BMI categories:
  (i) Healthy weight: 18.5 kg/m2 to 24.9 kg/m2 (ii) Overweight: 25 kg/m2 to 29.9 kg/m2 (iii) Obesity class 1: 30 kg/m2 to 34.9 kg/m2 (iv) Obesity class II: 35 kg/m2 to 39.9 kg/m2 (v) Obesity class III: ≥ 40 kg/m2
Proportion of Participants with change from baseline in waist-to-height ratio (WHtR ratio) categories at 48 weeks | 48 weeks
  Waist-to-height ratio WHtR ratio categories: <0.5; 0.5-0.59; ≥0.6.
Change from baseline in HbA1c (mmol/mol) at 48 weeks | 48 weeks
  To assess treatment effects on glucose metabolism and HbA1c.
Change from baseline at 48 weeks in Quality of Life Short Form 36 (SF-36) survey | 48 weeks
  Change from baseline at 48 weeks in Quality of Life Short Form 36 (SF-36) survey. To assess a subject's overall health related quality of life, as well as the physical functioning score. SF- 36 scores range from 0 (worst) to 100 (best).
Change from Baseline at 48 weeks in Impact of Weight on Quality of Life-Lite for Clinical Trials (IWQOL-Lite) | 48 weeks
  Change from baseline in IWQOL-Lite CT. IWQOL-Lite CT is a 20-item modified survey instrument that is used to quantitatively assess an individual's perception of how their weight affects their day- to-day life, as well as the physical function score. Scores range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Chair — Biomed Industries, Inc.
Locations (17):
- United States (8):
  - Biomed Research Unit #90067-102, Los Angeles, California
  - Biomed Research Unit # 92121-103, San Diego, California
  - Biomed Research Unit # 94104-101, San Francisco, California
  - Biomed Research Unit # 33012-104, Hialeah, Florida
  - Biomed Research Unit # 32256-105, Jacksonville, Florida
  - Biomed Research Unit # 33461-106, Lake Worth, Florida
  - Biomed Research Unit # 10021-107, New York, New York
  - Biomed Research Unit # 77479-108, Sugar Land, Texas
- Australia (5):
  - Biomed Research Unit-NSW-2100-109, Brookvale, New South Wales
  - Biomed Research Unit-NSW-2065-110, Saint Leonards,, New South Wales
  - , Australia, 4101 Biomed Research Unit-NSW-4101-111, South Brisbane, Queensland
  - Biomed Research Unit-VIC-3124-112, Camberwell, Victoria
  - , Victoria, Australia, 3084 Biomed Research Unit-VIC-3084-113, Heidelberg West, Victoria
- New Zealand (4):
  - Biomed Research Unit-NZ-1010-114, Auckland, Auckland
  - Biomed Research Unit-NZ-2025-115, Papatoetoe, Auckland
  - Hamilton, New Zealand, 3200 Biomed Research Unit-NZ-3200-116, Hamilton, New Zealand
  - Biomed Research Unit-NZ- 6242-117, Newtown, Wellington Region

IPD SHARING:
Plan to Share IPD: No